CLINICAL TRIAL: NCT04744948
Title: Effect Of Treadmill Based Aerobic Exercise Intervention On Menstruation And Quality Of Life In Women With Polycystic Ovarian Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Miral Saleh Mohamed, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETMQWP
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Polycystic Ovary Syndrome; Irregular Menses
MeSH Terms: conditions — Polycystic Ovary Syndrome; Menstruation Disturbances | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: control group receive low caloric diet study group receive high intensity interval training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low caloric diet (Placebo Comparator): low caloric diet 1200cal/day
  Interventions: Other: low caloric diet
- treadmill (Experimental): treadmill aerobic exercise training
  Interventions: Device: Treadmill exercise; Other: low caloric diet

INTERVENTIONS:
Device: Treadmill exercise — high intensity interval training
  Arms: treadmill
Other: low caloric diet — low caloric diet (1200ca/lday)

SUMMARY:
this study will be carried to investigate the effect of aerobic exercise on menstrual regularity and quality of life in pco women

DETAILED DESCRIPTION:
This study will be carried out on sixty females with polycystic ovarian syndrome (PCOS) patients will be randomly assigned into two equal groups: control group (30 women) will receive low caloric diet 1200 Cal/day) while study group (30 women) will receive the same diet regime and treadmill aeobic exercise

ELIGIBILITY:
Inclusion Criteria:

* women with pco
* age from17 to 28 years
* BMI 25- 30

Exclusion Criteria:

* Asthma and chronic respiratory disease
* congenital spinal problems
* cardiopulmonary disease
* physical impairments

Ages: 17 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — female hormones
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
menstrual regularity | 3 months
  Oligomenorrhea (menses every 6 weeks to 6 months), amenorrhea (menses greater than every 6 months apart or their absence), regular ( menses every 28-35 days)
quality of life questionnaire (QOLQ) | 3 months
  a total of 26 items for the Polycystic Ovary Syndrome Questionnaire, each question is associated with a 7-point scale in which 7 represents optimal function and 1 represents the poorest function

CONTACTS AND LOCATIONS:
Overall Officials: fahema m okiel, phd, Study Director — Cairo University; amal mo youssef, phd, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt